CLINICAL TRIAL: NCT00780377
Title: The Effects of Cardiac Innervation on Intra-coronary t-PA Release
Brief Title: Intracoronary Bradykinin Mediated t-PA Release in Heart Transplant Recipients
Acronym: P1A4D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to perform study due to unavailable drug, then unable to partner with cath lab
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 080823
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Heart Transplantation
Keywords: Heart Transplant; Fibrinolysis; Resting conditions
MeSH Terms: interventions — Bradykinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bradykinin (Experimental): Patients have holter monitoring. Patients receive intracoronary bradykinin (0.2, 0.6, 2.0 ug/min) and have coronary sinus and coronary artery blood sampling for t-PA and O2 content.
  Interventions: Drug: Bradykinin

INTERVENTIONS:
Drug: Bradykinin — Bradykinin 0, 0.2, 0.6, 2.0 ug/min intracoronary, for 5 minutes at each dose.

SUMMARY:
Heart transplant recipients do not have nerves to their hearts. This protocol tests the hypothesis that bradykinin mediated t-PA release in the coronary arteries will be reduced in heart transplant recipients compared to healthy subjects.

This study will compare heart transplant recipients to healthy controls who are undergoing cardiac cath for standard of care purposes (separate protocol) and compare the coronary arteries to the forearm in transplant recipients (separate protocol) and healthy controls (separate protocol).

ELIGIBILITY:
Inclusion criteria:

1. Heart transplant recipients undergoing annual cardiac catheterization who have participated our protocol: Characterization of brachial arterial t-PA release, vasodilator function, and vascular compliance and correlation with fibrinolytic balance, oxidative stress, and inflammation measures in heart transplant recipients (SCCOR Project 1, Aim 3C). (IRB # 070517)
2. 25 Subjects will have transplant vasculopathy and 25 subjects will be free of transplant vasculopathy, as documented in previous angiograms.
3. Otherwise healthy

Exclusion criteria:

1. PVC < 30
2. Hypertensive subjects on ACE inhibitors
3. Pregnant or nursing mothers
4. Diabetic with HbA1C > 7.5 or stigmata of end organ damage (neuropathy, retinopathy, nephropathy, cardiomyopathy)
5. Cholesterol > 30 mg/dL above NCEP accepted level based on cardiac risk.
6. Triglycerides > 200
7. Previously diagnosed obstructive coronary artery disease
8. Renal insufficiency (Creatinine ≥ 1.5 mg/dl)
9. History of cerebrovascular disease
10. Any chronic inflammatory disease (rheumatologic, inflammatory bowel disease, etc)
11. Uncontrolled Stage 2 Hypertension (160/100 mmHg), or end organ damage due to hypertension (left ventricular hypertrophy, atrial fibrillation, hematuria, renal insufficiency, prior cerebrovascular disease).
12. Angiotensin converting enzyme inhibitor use
13. Coagulopathy (INR ≥ 1.5, PTT ≥ 150% of control)
14. Peripheral Vascular Disease
15. Other chronic medical illnesses at the discretion of the investigators

Healthy controls are being enrolled in SCCOR Project 1, Aims 3A and 3B (IRB# 030473 and 061160) and will not be participating under this IRB number.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
T-PA release in the coronary artery bed. | Single Study Visit

SECONDARY OUTCOMES:
Heart rate variability | Single study visit
Histopathology for arteriolar t-PA and sympathetic neurons | Single Study Visit

CONTACTS AND LOCATIONS:
Overall Officials: James A S AS Muldowney, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States